CLINICAL TRIAL: NCT01531764
Title: Single-arm, Open-label, Multicentre Phase II Study Evaluating the Efficacy and Safety of BIBW 2992 (Afatinib) in Combination With Vinorelbine for the Treatment of Patients With Metastatic Breast Cancer With Intermediate HER2 Expression (HER2 2+ by Immunohistochemistry, Fluorescence In-situ Hybridisation (FISH) Negative) After Failure of First-line Therapy in the Metastatic Setting and Having Been Pre-treated With Anthracyclines
Brief Title: BIBW 2992 (Afatinib) and Vinorelbine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The recruitment was discontinued because of failure to meet expected enrolment goals
Sponsor: University of Magdeburg (Other)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.137
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2012-02

CONDITIONS: Carcinoma Breast Stage IV
Keywords: Metastatic breast cancer; intermediate HER2 expression; Afatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Afatinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: BIBW 2992 in combination with vinorelbine — Patients will receive BIBW 2992 and vinorelbine chemotherapy. BIBW 2992: 40 mg oral (tablet) once daily Vinorelbine: 25 mg/m² on days 1 & 8 in a 3-weekly course, intravenous, short infusion of about 10 minutes
  Other Names: Afatinib

SUMMARY:
This open-label, single-arm, multicentre phase II trial will be performed in patients with intermediate HER2-positive, metastatic breast cancer (MBC)pretreated with anthracyclines and one first-line therapy in the metastatic setting.

The main objective of the trial is to evaluate the efficacy and safety of BIBW 2992 in combination with vinorelbine in patients with intermediate HER2-positive MBC. If this trial shows promising results, further studies to evaluate the benefit of BIBW 2992 in combination with chemotherapy in this subgroup of intermediate HER2-positive patients with MBC are warranted.

Patients will be followed until progression. After progression, for the purpose of analysing overall survival, information on vital status and subsequent treatment will be collected.

The primary objective is to determine the 6-month progression free survival rate of BIBW 2992 and vinorelbine i.v. in patients with metastatic, HER2 IHC 2+, HER2 FISH-negative breast cancer.

BIBW 2992 in combination with vinorelbine will provide a suitable combination to test the hypothesis that patients with metastatic breast cancer whose tumours are HER2 2+ by immunohistochemistry, but negative by fluorescence in-situ hybridisation (FISH) will benefit from a combination of a cytotoxic agent, i.e. vinorelbine, plus the dual irreversible EGFR/HER2-tyrosine kinase inhibitor BIBW 2992.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years
* Histologically confirmed diagnosis of intermediate HER2-overexpressing breast cancer
* Stage IV metastatic disease
* Must have received anthracycline-based chemotherapy for adjuvant treatment of breast cancer or first-line treatment of metastatic breast cancer
* Must have received one first-line chemotherapy for metastatic breast cancer
* Must have (archived) tumour tissue sample available for central re- assessment of HER2 status and prove to be intermediate HER2-positive. HER2 intermediate status is defined as IHC 2+ and FISH-negativity.
* Must have at least one measurable lesion according to RECIST 1.1. Patient with only skin lesions will not be eligible.
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
* Life expectancy of at least six (6) months.
* Written informed consent that is consistent with ICH-GCP guidelines.
* Must be eligible for treatment with BIBW 2992 and vinorelbine.

Exclusion Criteria:

* 1. Prior treatment with EGFR/HER2-targeted tyrosine kinase inhibitors, i.e. lapatinib
* Prior treatment with vinorelbine
* Known pre-existing interstitial lung disease
* Radiotherapy, chemotherapy, hormone therapy, immunotherapy or surgery (other than biopsy) within 4 weeks (2 weeks for hormone therapy) prior to start of treatment with BIBW 2992 and vinorelbine.
* Active brain metastases
* Any other current malignancy or malignancy diagnosed within the past five (5) years (other than non-melanomatous skin cancer and in situ cervical cancer).
* Significant or recent acute gastrointestinal disorders with diarrhoea as a major symptom, e.g. Crohn's disease, malabsorption or CTC grade ≥ 2 diarrhoea of any aetiology.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of ≥3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to start of study treatment.
* Cardiac left ventricular function with resting ejection fraction of less than 50 %.
* Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
* Laboratory values according to specified ranges.
* Women of childbearing potential, unwilling to use a medically acceptable method of contraception during the trial.
* Pregnancy or breast-feeding.
* Patients unable to comply with the protocol.
* Known hepatitis B infection, known hepatitis C infection or known HIV carrier.
* Known or suspected active drug or alcohol abuse.
* Requirement for treatment with any of the prohibited concomitant medications
* Any contraindications for therapy with vinorelbine or BIBW 2992.
* Known hypersensitivity to BIBW 2992 or the excipients of any of the trial drugs.
* Use of any investigational drug within 4 weeks of start of treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival based on tumor imaging according to RECIST 1.1 criteria. | 6 months defined as the time from the date of treatment start
  The primary objective is to determine the 6-month Progression free survival rate of BIBW 2992 and vinorelbine i.v. in patients with metastatic, HER2 IHC 2+, HER2 FISH-negative breast cancer. The analysis will be based upon the evaluation of tumour imaging. Disease progression will be evaluated according to the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall survival including assessment of objective response rate and time to progression. | From start of treatment until the date of first documented progression or death from any cause, whichever came first, assessed approximately up to 24 months.
  Objective Response Rate based on Response Evaluation Criteria in Solid Tumours (RECIST 1.1), Time-to-Progression and Overall Survival.
Number, intensity and incidence of adverse events | Start of treatment up to 28 days after the last administration trial medication.
  Safety will be evaluated as indicated by number, intensity and incidence of adverse events, graded according to US NCI CTCAE Version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Bischoff, MD, Principal Investigator — Otto-von-Guericke-Universität Magdeburg, Germany
Locations (12):
- Germany (12):
  - Klinikum St. Marien Amberg, Amberg, Bavaria
  - Hämato-Onkologische Schwerpunktpraxis, München, Bavaria
  - Caritas-Krankenhaus, Onkologisches Zentrum Regensburg, Regenburg, Bavaria
  - Internistische Praxisgemeinschaft Eppendorf, Hamburg, Hamburg
  - OncoResearch Lerchenfled UG, Hamburg, Hamburg
  - Gynäkologische Praxis, Hildesheim, Lower Saxony
  - Schwerpunktpraxis für Hämatologie und Onkologie, Bottrop, North Rhine-Westphalia
  - Universitätsklinikum Frauenklinik Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Otto-von-Guericke-Universität Frauenklinik Magdeburg, Magdeburg, Saxony-Anhalt
  - Praxisklinik Krebsheilkunde für Frauen / Brustzentrum, Berlin, State of Berlin
  - Onkologisches Zentrum Süd, Vivantes Tumorzentrum, Berlin, State of Berlin